CLINICAL TRIAL: NCT06021041
Title: A Retrospective Study on the Treatment Pattern and Clinical Prognosis of Severe Tuberculosis Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Qin Ning, Professor, Tongji Hospital
Other Study IDs: RETUBO-S
Record Dates: First submitted 2023-08-21; First posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
This is a retrospective clinical study to analyze the clinical characteristics, complications, and effects of different treatment options on long-term prognosis of severe tuberculosis patients. All cases of severe tuberculosis diagnosed between 2016 and 2021 were included in the electronic medical record system of one center, and data such as demographics, hospitalization information, clinical information, laboratory or imaging examinations, treatment plans, and outcomes were collected.

ELIGIBILITY:
Inclusion Criteria:

1. For patients with severe pulmonary tuberculosis, imaging and grading diagnosis meet any of the following:

   1. Damaged lung ≥ 1 lobe
   2. Chest CT shows lesions in ≥3 lung lobes
   3. Hematogenous disseminated pulmonary tuberculosis
   4. caseous pneumonia
   5. bronchial tuberculosis
   6. Multiple hilar or mediastinal lymph node enlargement in primary pulmonary tuberculosis
   7. Rifampicin-resistant, multidrug-resistant, polydrug-resistant or pan-drug-resistant tuberculosis
   8. Combined more than 2 cavities over 8mm
   9. Tuberculous massive hemoptysis
   10. Pulmonary tuberculosis complicated with acute infection (including multidrug-resistant bacterial infection, fungal infection or multiple infection)
   11. Combined with extrapulmonary tuberculosis

       * Intracranial tuberculosis, spinal cord and/or meningeal tuberculosis
       * Pleural effusion, pericardial effusion

         * Empyema or empyema, hemopneumothorax, tracheobronchopleural fistula and severe infection.
         * Heart failure caused by cardiac tamponade or constrictive pericarditis
       * Multiple sites of lymphatic tuberculosis or surgery is necessary

         * Cervical lymphatic tuberculosis
         * Mediastinal lymphatic tuberculosis
         * Abdominal or retroperitoneal lymph node tuberculosis
       * Abdominal tuberculosis, tuberculous peritonitis (ascites or multiple serous cavities)

         * Intestinal tuberculosis causes complete or incomplete intestinal root obstruction or perforation or massive bleeding or severe abdominal infection
         * Gastrointestinal hemorrhage caused by tuberculosis of the digestive system, etc.
       * Musculoskeletal tuberculosis

         * Spinal (cervical, thoracic, lumbar, sacral) tuberculosis
         * Bones in other parts
         * Merge surrounding abscess
       * Urinary or renal tuberculosis

         * Renal failure or damaged blood vessels caused by renal tuberculosis
         * Ureteral stenosis or blockage caused by urinary tuberculosis
       * Adrenal tuberculosis in hypoadrenal insufficiency
       * Liver tuberculosis
2. Age and gender are not limited.

Exclusion Criteria:

* Patients with no clear diagnosis at discharge.
* Patients judged by the investigator to be unsuitable for inclusion in this protocol.
* The discharge diagnosis was central nervous system tuberculosis, or tuberculous meningitis, or tuberculous cerebrospinal meningitis, or tuberculous meningoencephalitis, or tuberculous encephalitis, or tuberculous brain abscess, or spinal tuberculosis, or tuberculous Hydrocephalus, and is currently participating in other clinical studies.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospitalized patients diagnosed with severe tuberculosis from the Grade A tertiary hospital in Hubei Province, China.
Sampling Method: Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2018-01-13 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
2-year survival rate | 2 years
  2-year survival rate
2-year disability rate | 2 years
  2-year disability rate

SECONDARY OUTCOMES:
The number of participants with the presence of clinical symptoms | 2 years
Incidence of complications in patients with different treatment regimens | 2 years
  Incidence of complications in patients with different treatment regimens
Length of hospital stay for patients | 2 years
  Length of hospital stay for patients
Proportion of patients admitted to the ICU | 2 years
  Proportion of patients admitted to the ICU

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Tongji Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Wuhan Pulmonary Hospital(Wuhan Institute for Tuberculosis Control), Hubei, Wuhan